CLINICAL TRIAL: NCT07088042
Title: "Assessment of Different Medications in Modifying the Efficacy of Anesthesia in Mandibular Molars With Acute Irreversible Pulpitis (A Randomized Clinical Trial)"
Brief Title: Assessment of Different Medications in Modifying the Efficacy of Anesthesia in Mandibular Molars With Acute Irreversible Pulpitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FDASU-RecIM012370
Record Dates: First submitted 2025-05-06; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: Pulpitis - Irreversible
Keywords: premedication; bromelain trypsin chymotrypsin; efficacy of anesthesia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Non-Steroidal Anti-inflammatory drug (Cataflam 50mg) (Active Comparator): Received Cataflam
  Interventions: Drug: Cataflam® 50 coated tablet
- Inferior alveolar nerve block only (No Intervention): received Inferior alveolar nerve block only
- Oral Tablets of Limitless Allzyme (Experimental)
  Interventions: Drug: Limitless Allzyme
- Alphintern® (Trypsin/Chymotrypsin 5 micro Katals/14 micro Katals) (Active Comparator)
  Interventions: Drug: Oral tablets of Alphintern®

INTERVENTIONS:
Drug: Limitless Allzyme — Received Limitless Allzyme Max® Trypsin/Chymotrypsin/Bromelain(15 microkatal/42microkatal/240 GDU)
  Arms: Oral Tablets of Limitless Allzyme
Drug: Oral tablets of Alphintern® — received (Trypsin/Chymotrypsin 5 micro Katals/14 micro Katals)
  Arms: Alphintern® (Trypsin/Chymotrypsin 5 micro Katals/14 micro Katals)
Drug: Cataflam® 50 coated tablet — of Cataflam 50 mg as part of their treatment protocol
  Arms: Non-Steroidal Anti-inflammatory drug (Cataflam 50mg)

SUMMARY:
The goal of this clinical trial is to assess the effect of preoperative

* Oral Tablets of Trypsin/Chymotrypsin/Bromelain Limitless Allzyme® (15 microkatal/42microkatal/240 GDU)
* Oral tablets of Alphintern® (Trypsin/Chymotrypsin 5 micro Katals/14 micro Katals)
* Oral Tablets Non-Steroidal Anti-inflammatory drug (Cataflam® 50mg)

Regarding the efficacy of the inferior alveolar nerve block anesthesia in mandibular molars with symptomatic irreversible pulpitis and post operative pain follow up for 3 days.

The main question it aims to answer are: • Does premedication increase the success rate of inferior alveolar nerve block.

Participants will describe their preoperative pain level to the investigator and describe their pain level during the treatment. Researchers will compare different premedication to see if it increases the success rate of inferior alveolar nerve block using Visual Analogue Scale (VAS), Electric Pulp testing and cavity test.

ELIGIBILITY:
Inclusion Criteria:

* • From 18 to 65 years old.

  * Both male and female participants were accepted.
  * Mandibular molars diagnosed with acute irreversible pulpitis.
  * Class I occlusion with normal occlusal contacts

Exclusion Criteria:

* • Individuals with significant health issues: a history of gastrointestinal disorders, active bronchial asthma, renal diseases, liver dysfunction, heart diseases, blood disorders, hypertension or poorly controlled diabetes mellitus.

  * Immunocompromised patients.
  * Sensitivity or allergy to any of the pharmaceuticals or medications intended for use in the study
  * Participants who could not read, comprehend, or complete the baseline pain scale questionnaire.
  * Cases where clinical examination suggested necrotic teeth leading to a false positive diagnosis.
  * Teeth exhibiting periodontal disease or periapical lesions confirmed through clinical assessment and pre-operative radiographs.
  * Sensitivity to percussion or palpation in the included teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
assess the effect of Preoperative administration of- Oral tablets of Trypsin/Chymotrypsin/Bromelain) - Regarding the efficacy of the inferior alveolar nerve block anesthesia in mandibular molars with symptomatic irreversible pulpitis | Up to 30 minutes from lip numbness until the end of pulp exacerbation and post operative pain follow up for 3 days.
  Assessment of outcome is done using cavity test.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hashem AAR, Abd El Sattar AA, Abdel Rahman TY. The Effect of Trypsin-Chymotrypsin on Postoperative Pain after Single Visit Endodontic Treatment: A Randomized Controlled Trial. J Endod. 2023 Mar;49(3):240-247. doi: 10.1016/j.joen.2022.12.010. Epub 2022 Dec 24. PMID 36574828